CLINICAL TRIAL: NCT05480774
Title: The Assessment for Effect of Red Ginseng Extract on Changes in Indicators of Immune Function in Vietnamese Healthy Volunteers: The Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Effect of Red Ginseng Extract on Changes in Indicators of Immune Function in Vietnamese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre of Clinical Pharmacology, Hanoi Medical University (Other)
Collaborators: Kyunghee University (Other); HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BMRI-CT-2021-01
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KRG hard capsules (Active Comparator): Each KRG hard capsule contains 500 mg of red ginseng extract. Dosage of KRG hard capsule: oral administration of 1 capsule twice daily for 12 weeks.
  Interventions: Drug: KRG hard capsule
- Placebo hard capsules (Placebo Comparator): The composition of the Placebo hard capsule contains red ginseng flavor. Dosage of Placebo hard capsule: oral administration of 1 capsule twice daily for 12 weeks.
  Interventions: Drug: Placebo hard capsule

INTERVENTIONS:
Drug: KRG hard capsule — Each subject was given orally 2 KRG hard capsules/day for 12 weeks
  Arms: KRG hard capsules
Drug: Placebo hard capsule — Each subject was given orally 2 placebo hard capsules/day for 12 weeks
  Arms: Placebo hard capsules

SUMMARY:
This is a placebo-controlled, randomized, double-blind, multiple dose study that evaluated the safety, tolerability, and changes in indicators of immune function of Korean Red Ginseng Extract in Vietnamese healthy subjects following oral administration of multiple dose of Korean Red Ginseng Extract as hard capsules or placebo to healthy adult men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female aged 20 to 65 years, inclusive at the time of informed consent
* Have not any abnormalities of vital signs (temperature, systolic blood pressure (SBP) and diastolic blood pressure (DBP) and pulse rate), physical examinations, clinical laboratory tests (hematology, chemistry, and urinalysis).
* Ability and willingness to provide written informed consent and to comply with the requirements of the protocol.
* Peripheral white blood cells in the range of 3000 - 10,000/μL
* Subjects with a history of being infected with COVID-19 within 12 months according to the diagnostic criteria of the Ministry of Health at the time of infection

Exclusion Criteria:

* Pregnancy or lactation
* For subjects of reproductive potential, a positive result from a serum pregnancy test at screening, or not willing to use reliable means of contraception
* Evidence of clinically significant acute or chronic hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psych, neurological, or neoplastic diseases (however, at the discretion of the principal investigator, subjects may also be considered)
* Uncontrolled hypertension (SBP ≥160 mmHg and/or DBP ≥100 mmHg, measured following at least 10 mins of rest)
* Uncontrolled diabetes (fasting glucose level above 126 mg/dL or diabetic patients who have initial treatment with antidiabetic drugs for ≤ 3 months)
* Aspartate aminotransferase or alanine aminotransferase >=3.0 × upper limit of normal
* Serum creatinine level > 2,4 mg/dL for male and > 1,8 mg/dL for female
* Use of medications and dietary supplements that can affect immunity within 2 weeks before screening
* Those who complain of severe gastrointestinal symptoms such as heartburn and indigestion
* History of sensitivity or allergy to investigational product-related foods
* Plan to participate in other research while participating in this research
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study.
* Failure of follow instructions for discontinuing immune-affecting dietary supplements during the wash-out period prior to trial participation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with the administration of KRG | 12 weeks
  Frequency and characteristics of adverse events associated with the administration of KRG

SECONDARY OUTCOMES:
Natural killer (NK) cell count | 12 weeks
  Change in NK cell count after 12 weeks compared to baseline
White blood cell count | 12 weeks
  Change in white blood cell count after 12 weeks compared to baseline
Interferon (IFN)-α, β, γ levels | 12 weeks
  Changes in IFN-α, β, γ levels after 12 weeks compared to baseline
Tumor necrosis factor (TNF)-α, β, γ levels | 12 weeks
  Changes in TNF-α, β, γ levels after 12 weeks compared to baseline
Interleukin (IL)-1, 4, 6 levels | 12 weeks
  Changes in IL-1, 4, 6 levels after 12 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Clinical Pharmacology, Hanoi, Vietnam